CLINICAL TRIAL: NCT06520124
Title: Effectiveness of Essilor® Stellest® Lenses in Slowing Down Myopia Progression in Young Adults
Brief Title: Stellest Lens Wear in Adult Progressing Myopes
Acronym: SWAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FCBMS-24-022
Record Dates: First submitted 2024-07-09; First posted 2024-07-25 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-07

CONDITIONS: Myopia, Progressive
Keywords: Adult myopia; Progressing adult myopes; Stellest; HAL; Progressive myopia; Myopia; Refractive error; Axial length
MeSH Terms: conditions — Myopia, Degenerative; Myopia; Refractive Errors

STUDY DESIGN:
Intervention Model Description: Participants will wear the treatment lens in front of one eye and a single vision lens in front of the other eye (Arms A1 and A2). This will be randomised by eye dominancy and crossed-over after one year (Arms B1 and B2).
Masking Description: Not possible to mask as participant and/or investigator could identify which lens is 'different' from single-vision through visual inspection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (4):
- A1: Stellest lens wear in front of dominant eye (Experimental): Stellest lens wear in front of dominant eye.
  Interventions: Device: Essilor® Stellest® spectacle lens
- A2: Single vision lens wear in front of non-dominant eye (Placebo Comparator): Single vision lens wear in front of non-dominant eye.
  Interventions: Device: Single-vision spectacle lens
- B1: Stellest lens wear in front of non-dominant eye (Experimental): Single vision lens wear in front of non-dominant eye
  Interventions: Device: Essilor® Stellest® spectacle lens
- B2: Single-vision lens wear in front of dominant eye. (Placebo Comparator): Single vision lens wear in front of dominant eye.
  Interventions: Device: Single-vision spectacle lens

INTERVENTIONS:
Device: Essilor® Stellest® spectacle lens — Spectacle lens with highly aspherical lenslets.
  Other Names: Highly Aspherical Lenslets; HAL; Stellest; Essilor Stellest; HALT
  Arms: A1: Stellest lens wear in front of dominant eye; B1: Stellest lens wear in front of non-dominant eye
Device: Single-vision spectacle lens — Standard single-vision distance spectacle lens.
  Other Names: Single-vision lens; single vision lens
  Arms: A2: Single vision lens wear in front of non-dominant eye; B2: Single-vision lens wear in front of dominant eye.

SUMMARY:
It is expected that myopia progression stabilises in the late teenage years, however, some studies report that myopia progression continues through early adulthood in as many as one third of myopes. Similarly, there are reports of myopia commencing in early adulthood. Although the rate of progression is slower than that occurring in childhood, between 20-35% of adults aged between 20-30 years were reported to progress by at least -1.00D over a five year period. Given that every dioptre increase in myopia results in an increased overall lifetime risk of serious ocular pathology, it seems opportune to investigate whether myopia management treatments designed to slow myopia progression in childhood could be beneficial for progressing adult myopes. The proposed study will conduct a prospective, randomised, paired-eye, trial with cross-over to evaluate the efficacy of Essilor Stellest myopia management spectacle lenses on the progression of myopia in adults aged between 18-40 years. The outcomes from the trial will provide novel evidence regarding the utility of these lenses in an adult population.

DETAILED DESCRIPTION:
This is a 2-year, prospective, randomised, paired-eye controlled trial with cross-over which will be conducted at Ulster University, Coleraine, Northern Ireland. The trial will evaluate the efficacy of Essilor Stellest myopia management spectacle lenses on the progression of myopia in adults aged between 18-40 years. Participants will act as their own control, wearing a Stellest lens in front of one eye and a single vision lens in front of the fellow eye. At the 12-month visit, lens allocation will be crossed-over between eyes and worn for a further 12 months. Randomisation of whether Stellest will be worn in the dominant or non-dominant eye first will be conducted using permuted block design.

Participants will be asked to wear the study spectacles for at least 12 hours per day, 6 days per week. No other form of myopia management spectacle or contact lens will be worn during the trial period. At the two-year review participants will be given the option of continuing with Stellest lenses in both eyes or reverting to single vision spectacles in both eyes depending on the results of the study. Those participants who continue to wear Stellest lenses (binocularly) will be contacted after one month to investigate the acceptability of Stellest wear in adult myopes.

Participants will be screened at baseline to ensure they meet the inclusion criteria. Participants will be asked if they have ever attended the hospital eye service or have been told they have an eye condition by their optometrists. Fundus images and slit lamp examination will also be conducted at baseline to confirm eye health. Cycloplegic refraction and axial length will be measured at baseline, 6-months and 12-months using the Shin-Nippon NVision-K 5001 and IOLMaster 700 respectively. Cycloplegia will be induced by two drops of 1% tropicamide separated by 5 minutes. Punctal occlusion following instillation of the drop will be applied to reduce systemic absorption.

At 12-months, the crossover will take place. A further assessment of cycloplegic refraction and axial length will be performed 6-months (18-month visit) and 12-months (24-month visit) after the crossover. The following additional measurements will also be made to inform parameters that are associated with better response to treatment and to ensure visual function remains adequate while wearing the study spectacles. These measurements will be taken at baseline and crossover.

* Near and distance visual acuity will be measured using a crowded logMAR letter chart at 33cm and 3m
* Accommodative function will be assessed using dynamic retinoscopy using the UC-Cube
* Binocularity will be assessed using distance and near prism cover test
* Field of vision will be assessed using a Humphrey suprathreshold screening test
* Peripheral refraction will be measured at 30 degrees nasally and temporally
* Choroidal thickness will be measured using a six radial scan using the Heidelberg Spectralis
* Visual comfort will be surveyed by telephone one week after collection of the study spectacles to ensure participants are tolerating the paired-eye control condition

ELIGIBILITY:
Inclusion Criteria:

* Cycloplegic SER less than -0.75D
* Astigmatism of 1.50D or less
* Anisometropia of 1.50D or less
* Evidence of annual progression of myopia of at least 0.50D in the previous two-year period

Exclusion Criteria:

* Previous myopia management (other than standard spectacle or contact lens correction)
* Ocular and systemic diseases which might affect visual performance or myopia development

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in axial length (mm) | 2 years
  Change in axial length (mm) of the eye wearing the Stellest lens compared to the control eye wearing standard single vision lenses.
Change in cycloplegic autorefraction (D) | 2 years
  Change in cycloplegic autorefraction (D) of the eye wearing the Stellest lens compared to the control eye wearing standard single vision lenses.

SECONDARY OUTCOMES:
Acceptability to adult patients of Stellest lenses prescribed for both eyes, assessed using the Stellest adult tolerability questionnaire. | 1 month
  Acceptability to adult patients of the Stellest lens when prescribed for both eyes following the 2-year trial period.

CONTACTS AND LOCATIONS:
Overall Officials: Sara J McCullough, PhD, Principal Investigator — Ulster University
Locations (1):
- Ulster University, Coleraine, County Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data.

REFERENCES:
- [Background] Stern E. Cytohistopathology of cervical cancer. Cancer Res. 1973 Jun;33(6):1368-78. No abstract available. PMID 4718680
- [Background] Bullimore MA, Reuter KS, Jones LA, Mitchell GL, Zoz J, Rah MJ. The Study of Progression of Adult Nearsightedness (SPAN): design and baseline characteristics. Optom Vis Sci. 2006 Aug;83(8):594-604. doi: 10.1097/01.opx.0000230274.42843.28. PMID 16909085
- [Background] Parssinen O, Kauppinen M, Viljanen A. The progression of myopia from its onset at age 8-12 to adulthood and the influence of heredity and external factors on myopic progression. A 23-year follow-up study. Acta Ophthalmol. 2014 Dec;92(8):730-9. doi: 10.1111/aos.12387. Epub 2014 Mar 27. PMID 24674576
- [Background] Lee SS, Lingham G, Sanfilippo PG, Hammond CJ, Saw SM, Guggenheim JA, Yazar S, Mackey DA. Incidence and Progression of Myopia in Early Adulthood. JAMA Ophthalmol. 2022 Feb 1;140(2):162-169. doi: 10.1001/jamaophthalmol.2021.5067. PMID 34989764
- [Background] Flitcroft DI. The complex interactions of retinal, optical and environmental factors in myopia aetiology. Prog Retin Eye Res. 2012 Nov;31(6):622-60. doi: 10.1016/j.preteyeres.2012.06.004. Epub 2012 Jul 4. PMID 22772022
- [Background] Anstice NS, Phillips JR. Effect of dual-focus soft contact lens wear on axial myopia progression in children. Ophthalmology. 2011 Jun;118(6):1152-61. doi: 10.1016/j.ophtha.2010.10.035. Epub 2011 Jan 26. PMID 21276616
- [Background] McCullough S, Adamson G, Breslin KMM, McClelland JF, Doyle L, Saunders KJ. Axial growth and refractive change in white European children and young adults: predictive factors for myopia. Sci Rep. 2020 Sep 16;10(1):15189. doi: 10.1038/s41598-020-72240-y. PMID 32938970
- [Background] Bao J, Huang Y, Li X, Yang A, Zhou F, Wu J, Wang C, Li Y, Lim EW, Spiegel DP, Drobe B, Chen H. Spectacle Lenses With Aspherical Lenslets for Myopia Control vs Single-Vision Spectacle Lenses: A Randomized Clinical Trial. JAMA Ophthalmol. 2022 May 1;140(5):472-478. doi: 10.1001/jamaophthalmol.2022.0401. PMID 35357402